CLINICAL TRIAL: NCT06321744
Title: Study Evaluating the Feasibility of an Adapted Physical Activity Program During the Hospitalization Phase in Cancer Patients Undergoing Treatment
Acronym: PREVAPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/825
Record Dates: First submitted 2024-03-07; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: Physical exercise; cancer; hospitalization
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted physical activity program (APA Program) (Experimental): An intervention (APA program) will be offered to patients hospitalized in the conventional hospitalization department of the medical oncology department.
  At entry, after presenting the study and obtaining non-opposition from patients, an initial assessment will be carried out before the APA program.
  At the end of the initial assessment, an APA program supervised (individually and in a room) by an APA teacher will be offered to patients. The sessions will be offered daily to patients (maximum 5 times/week). They will last on average 20 minutes each depending on the fatigue, pain and fitness of the patients. The objectives pursued are mainly an improvement in functional independence and mobility.
  Interventions: Other: adapted physical activity program (APA Program)

INTERVENTIONS:
Other: adapted physical activity program (APA Program) — Content of the APA program:
  * Strengthening of the lower limbs: Exercises alternating different regimes of muscular contractions (eccentric, concentric and isometric), with the use of elastics, balls or even body weight. These exercises will mainly work the quadriceps and hamstrings.
  * Upper limb strengthening: Exercises focused on eccentric and concentric contraction regimes, in a global movement approach (as opposed to a segmental approach), with the use of elastics, dumbbells, weighted balls, etc. These exercises will work the muscles of the biceps, triceps, pectorals, deltoids and lats.
  * Walking: In the room and/or in the corridor, with technical assistance (cane/walker, etc.) or human work
  * Balance and proprioception: Balance work in a bi- and uni-pedal situation, statically and dynamically (eyes open and closed) will be offered with the use of proprioception boards and/or mats combining if possible work in dual task.

SUMMARY:
This is a non-randomized, non-controlled feasibility study which will take place at the Besançon University Hospital in the conventional hospitalization department.

It will be carried out with patients hospitalized in the conventional hospitalization department of the medical oncology department of Besançon University Hospital.

At entry, after presenting the study and obtaining non-opposition from patients, an initial assessment will be carried out before the APA program. This assessment will include an evaluation of physical parameters (measurements of body composition, functional capacities, autonomy in activities of daily living and muscular strength), as well as an evaluation of quality of life relating to health and motivation to practice physical activity.

At the end of the initial assessment, an APA program supervised (individually and in a room) by an APA teacher will be offered to patients. The sessions will be offered daily to patients (maximum 5 times/week). They will last on average 20 minutes each depending on the fatigue, pain and fitness of the patients. The objectives pursued are mainly an improvement in functional independence and mobility.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 and over (no age limit)
* Patient followed for cancer,
* Patients with no medical contraindication to adapted physical activity (certificate)
* Patient with a performance index status less than 4
* Patient hospitalized in the conventional medical oncology hospitalization department of Besançon University Hospital.
* Patient not opposed to participating in the study
* Patient affiliated to a French social security scheme or beneficiary of such a scheme.
* For women: menopausal for at least 24 months, surgically sterilized, or, for women of childbearing age, use an effective method of contraception (oral contraceptives, contraceptive injections, intrauterine devices, double-barrier method, patches contraceptives)
* Length of hospitalization estimated at at least 7 days (main objective) and with the patient's objective of returning home or to SSR in the long term

Exclusion Criteria:

* Patient with an absolute medical contraindication to adapted physical activity
* Patient with inability to understand instructions and complete questionnaires.
* Patient with a performance index status of 4
* Patient with legal incapacity or limited legal capacity
* Patient unlikely to cooperate in the study and/or low cooperation anticipated by the investigator
* Patient without health insurance
* Pregnant woman
* Patient being in the exclusion period of another study or provided for by the "national volunteer file".

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Validate the feasibility of a supervised adapted physical activity (APA) program during the first 7 days of hospitalization in medical oncology for patients with cancer undergoing treatment | 7 days after inclusion
  The main objective of the study is to validate that the proportion of patients having completed, from inclusion (D0), at least three supervised APA sessions of a minimum duration of 15 minutes, during the first 7 consecutive days of his hospitalization (P) is beyond a threshold considered uninteresting of 50% (P0)
  To test the following hypotheses:
  H0: a compliant patient rate <= 50% is uninteresting (P<=P0) H1: a compliant patient rate > 80% is expected (P>P1) With an A'Hern type design, a one-sided alpha risk of 2.5% and a power of 90%, it is required to include 28 evaluable patients in the study to test H0 vs H1.
  Considering a rate of unevaluable patients of 10% it will be necessary to include 32 patients.
  Hypothesis H0 will be rejected if 20 (71.4%) or more than 20 patients out of the first 28 evaluable are compliant.

SECONDARY OUTCOMES:
Describe the evolution of body composition measured by impedancemetry | At inclusion (day 1) and at the study completion, an average of 15 days
  * fat-free mass index and muscle mass,
  * body protein content,
  * metabolic activity index
Describe the evolution of physical parameters functional capacities | At inclusion (day 1) and at the study completion, an average of 15 days
  - Score of Short Physical Performance Battery Test (Score of 0 =Faible performance to 12= Haute performance)
Describe the evolution of autonomy in daily life activities | At inclusion (day 1) and at the study completion, an average of 15 days
  IADL Questionnaire IADL score 0 to 4
  * IADL score = 0: dependent
  * IADL score = 4 autonomous
Describe the evolution of muscular strength | At inclusion (day 1) and at the study completion, an average of 15 days
  Handgrip :results in kilograms
Describe the evolution of the quality of life | At inclusion (day 1) and at the study completion, an average of 15 days
  QLQ-C30 questionnaire All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Describe the evolution of motivation to practice physical activity | At inclusion (day 1) and at the study completion, an average of 15 days
  Questionnaire BREQ-2 The BREQ-2 is a 19 item questionnaire that measures the stages of the self-determination continuum with respect to motivation to exercise with a 5 point Likert scale (0=not true for me, 4=very true for me)
Tolerance with the APA program on perception of effort | immediately after each intervention session
  Perception of effort with te Borg scale CR10.
  Scale of 0 (No exertion at all) to 10 (representing an extreme intensity of activity)
Tolerance with the APA program on pain and fatigue | Immediately before and after each intervention session
  Visual analog scale (0 = no pain and 10 = very severe pain)
Tolerance with the APA program on fatigue | Immediately before and after each intervention session
  Visual analog scale (0 = no fatigue and 10 = very severe fatigue)
Compliance with the APA program | at the study completion, an average of 15 days
  Number of sessions carried out out of the number planned
Criteria/reasons for non-participation, non-compliance, discontinuation of the intervention and study withdrawals | at the study completion, an average of 15 days
Patient satisfaction | at the study completion, an average of 15 days
  Likert scale (0= unsatisfiedt o 5 =very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Quentin JACQUINOT, Dr, Principal Investigator — CHU Besançon

IPD SHARING:
Plan to Share IPD: No